CLINICAL TRIAL: NCT05361070
Title: Neonatal Seizure Registry, GEnetics of Post-Neonatal Epilepsy (NSR-GENE)
Brief Title: Neonatal Seizure Registry, GEnetics of Post-Neonatal Epilepsy
Acronym: NSR-GENE
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-35563; R01NS124051 (NIH); R01NS124051-01A1 (NIH)
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Neonatal Seizure; Hypoxic-Ischemic Encephalopathy; Stroke; Intracranial Hemorrhage; Epilepsy; Gene Abnormality
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Stroke; Intracranial Hemorrhages; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: None Retained — Saliva and buccal swab for DNA extraction
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The NSR-GENE study is a longitudinal cohort study of approximately 300 parent-child trios from the Neonatal Seizure Registry and participating site outpatient clinics that aims to evaluate whether and how genes alter the risk of post-neonatal epilepsy among children with acute provoked neonatal seizures. The researchers aim to develop prediction rules to stratify neonates into low, medium, and high risk for post-neonatal epilepsy based on clinical, electroencephalogram (EEG), magnetic resonance imaging (MRI), and genetic risk factors.

DETAILED DESCRIPTION:
Neonatal seizures due to brain injury (acute provoked seizures) are associated with high risk of post-neonatal epilepsy. Although clinical risk factors can help predict which children are at highest risk for epilepsy, little is known about how genetic factors modify the risk for epilepsy after acute provoked neonatal seizures. The Neonatal Seizure Registry - GENetics of Epilepsy (NSR-GENE) study will test the central hypothesis that children who develop post-neonatal epilepsy are more likely to have pathogenic variants in epilepsy genes, and enrichment in single nucleotide polymorphisms within key inflammatory, neurotransmitter transport and homeostasis, and neurotrophic gene pathways as compared with children who do not develop unprovoked seizures before age five years, and that these can be added to traditional clinical risk factors to predict epilepsy after neonatal seizures.

ELIGIBILITY:
Inclusion Criteria:

* Children < 44 weeks postmenstrual age at seizure onset
* Seizures due to an acute provoked cause (including, but not limited to HIE, ischemic stroke, or intracranial hemorrhage)
* Parent(s) who are English or Spanish literate (with interpreter)
* Birthdate between 3/1/2023 and 1/1/2011
* One biological parent willing to participate
* Enrolled in NSR-II
* Fulfilling all NSR-II eligibility criteria and evaluated at an NSR center for neonatal seizures or enrolled in NSR-RISE

Exclusion Criteria:

* Risk for adverse outcome independent of seizures and underlying brain injury (including but not limited to inborn errors of metabolism, fetal infection, brain malformation)
* Transient cause for seizures (e.g., hypoglycemia without brain injury, hyponatremia, hypocalcemia)
* Neonatal-onset epilepsy syndromes
* Deceased

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient, family members/caregivers, children/minors, participants unable to read, speak or understand English
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with post-neonatal epilepsy | 5 years of age
  The presence or absence of a post-neonatal epilepsy diagnosis at age 5 in children with a prior history of acute symptomatic neonatal seizures will be determined by telephone interview with the parent and corroborated by medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Hannah C Glass, MDCM, MAS, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
In accordance with study sponsor
Time Frame: In accordance with study sponsor
Access Criteria: In accordance with study sponsor

REFERENCES:
- [Background] Shellhaas RA, Wusthoff CJ, Numis AL, Chu CJ, Massey SL, Abend NS, Soul JS, Chang T, Lemmon ME, Thomas C, McNamara NA, Guillet R, Franck LS, Sturza J, McCulloch CE, Glass HC. Early-life epilepsy after acute symptomatic neonatal seizures: A prospective multicenter study. Epilepsia. 2021 Aug;62(8):1871-1882. doi: 10.1111/epi.16978. Epub 2021 Jul 2. PMID 34212365
- [Background] Numis AL, da Gente G, Sherr EH, Glass HC. Whole-exome sequencing with targeted analysis and epilepsy after acute symptomatic neonatal seizures. Pediatr Res. 2022 Mar;91(4):896-902. doi: 10.1038/s41390-021-01509-3. Epub 2021 Apr 12. PMID 33846556
- [Background] Glass HC, Grinspan ZM, Li Y, McNamara NA, Chang T, Chu CJ, Massey SL, Abend NS, Lemmon ME, Thomas C, McCulloch CE, Shellhaas RA; Neonatal Seizure Registry Study Group. Risk for infantile spasms after acute symptomatic neonatal seizures. Epilepsia. 2020 Dec;61(12):2774-2784. doi: 10.1111/epi.16749. Epub 2020 Nov 13. PMID 33188528
- [Background] Glass HC, Grinspan ZM, Shellhaas RA. Outcomes after acute symptomatic seizures in neonates. Semin Fetal Neonatal Med. 2018 Jun;23(3):218-222. doi: 10.1016/j.siny.2018.02.001. Epub 2018 Feb 6. PMID 29454756
- [Background] Bennett ER, Reuter-Rice K, Laskowitz DT. Genetic Influences in Traumatic Brain Injury. In: Laskowitz D, Grant G, editors. Translational Research in Traumatic Brain Injury. Boca Raton (FL): CRC Press/Taylor and Francis Group; 2016. Chapter 9. Available from http://www.ncbi.nlm.nih.gov/books/NBK326717/ PMID 26583176
- [Background] Wong VS, Langley B. Epigenetic changes following traumatic brain injury and their implications for outcome, recovery and therapy. Neurosci Lett. 2016 Jun 20;625:26-33. doi: 10.1016/j.neulet.2016.04.009. Epub 2016 May 4. PMID 27155457
- [Background] Christensen J, Pedersen MG, Pedersen CB, Sidenius P, Olsen J, Vestergaard M. Long-term risk of epilepsy after traumatic brain injury in children and young adults: a population-based cohort study. Lancet. 2009 Mar 28;373(9669):1105-10. doi: 10.1016/S0140-6736(09)60214-2. Epub 2009 Feb 21. PMID 19233461
- [Background] Eriksson H, Wirdefeldt K, Asberg S, Zelano J. Family history increases the risk of late seizures after stroke. Neurology. 2019 Nov 19;93(21):e1964-e1970. doi: 10.1212/WNL.0000000000008522. Epub 2019 Oct 23. PMID 31645466